CLINICAL TRIAL: NCT06362018
Title: A Comparative Pharmacokinetic Profiles of Five Urolithin A Formulations in Healthy Volunteers: A Randomized, Open-label, Single-dose, Parallel-arm Study
Brief Title: Bioavailability of Five Mitopure Formulations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Collaborators: Mprex Healthcare Pvt. Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MHC/CT/23-24/055; MHC/CT/23-24/055, Version No.: (Other: Mprex Healthcare Pvt. Ltd.)
Record Dates: First submitted 2024-04-02; First posted 2024-04-12 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Healthy Adults
Keywords: Mitopure; Urolithin A; Bioavailability
MeSH Terms: interventions — 3,8-dihydroxy-6H-dibenzo(b,d)pyran-6-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Formulation A (Active Comparator)
  Interventions: Dietary Supplement: Mitopure (Urolithin A)
- Formulation B (Experimental)
  Interventions: Dietary Supplement: Mitopure (Urolithin A)
- Formulation C (Experimental)
  Interventions: Dietary Supplement: Mitopure (Urolithin A)
- Formulation D (Experimental)
  Interventions: Dietary Supplement: Mitopure (Urolithin A)
- Formulation E (Experimental)
  Interventions: Dietary Supplement: Mitopure (Urolithin A)

INTERVENTIONS:
Dietary Supplement: Mitopure (Urolithin A) — Mitopure (Urolithin A) is gut microbiome derived postbiotic that has been shown to improve muscle and mitochondrial health

SUMMARY:
This study's design as an open-label, single-dose, randomized trial that aligns with the objective of characterizing the concentration-time profiles of five Urolithin A (Mitopure) formulations in a controlled setting. The inclusion criteria, stringent fasting requirements, standardized fluid intake and strict dietary restriction protocols ensure homogeneity among the study participants, enhancing the reliability of the outcomes.

Ultimately, this clinical trial aims to contribute valuable insights into the pharmacokinetic behavior of the different Urolithin A formulations, facilitating informed decisions for future developments and applications in the realm of health and wellness.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female participants aged between 18 and 45 years (both inclusive);
2. Non-smoker subject or smoker of not more than 5 cigarettes a day;
3. Body Mass Index (BMI) between 18.50-30.00 kg/m2 inclusive;
4. Trial participants in normal health as determined by personal medical history, clinical examination including vital signs, and clinically acceptable results of laboratory examinations (including serological tests), individual values out of the normal range can be accepted if judged clinically non relevant by the Investigator;
5. Normal ECG recording on a 12-lead ECG and/or chest X-ray (PA view) significant at the screening visit or considered not clinically significant (NCS) by investigators;
6. A negative alcohol breath test result at housing;
7. Trial participant able to communicate effectively, provide voluntary written informed consent and available for the entire study duration;
8. Trial participants willing to adhere to the protocol requirements as evidenced by written informed consent approved by the ethics committee;
9. Ability to fast for at least 14.00 hours and consume standard meals;
10. Accept to refrain consuming certain foods and supplements at least two weeks before inclusion;
11. Female participants must have a negative urine pregnancy test prior to housing; 12.Trial participants that can provide adequate evidence of their identity;

13.The participants agree to refrain from consuming dietary supplements that could potentially impact either muscle or mitochondrial function or contain Urolithin A, such as resveratrol, pomegranate and ellagitannins, nicotinamide riboside, whey protein, leucine, iso-leucine, l-carnitine, creatinine, coenzyme Q10, vitamin A, niacin, folic acids, vitamin C, vitamin E and probiotic foods and supplements, during the 2 weeks before inclusion and throughout the study; 14.Females of childbearing potential agree to use appropriate contraceptive measures like non-hormonal intrauterine devices, barrier methods, and spermicidal agents during the study and 07 days after completion of the study; 15.Male agreeing to use appropriate contraceptive measures like the Double Barrier method (Condom), and should not donate sperm, etc. during the study and 07 days after completion of the study.

Exclusion Criteria:

1. Known hypersensitivity to Urolithin A or related product or any component of intervention, presence or history of drug hypersensitivity, allergic disease or lactose intolerance;
2. Any history or presence of clinically significant medical condition, such as, but not limited to, cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, hematological, neurologic, psychiatric, systemic or infectious disease, thyroid disease, adrenal dysfunction, or organic intracranial lesion;
3. Any treatment which could bring about induction or inhibition of the hepatic microsomal enzyme system within one month of starting the study;
4. History or presence of alcoholism or drug abuse;
5. History or presence of gastric and/or duodenal ulceration;
6. History or presence of cancer;
7. Difficulty with donating blood;
8. Use of any prescribed medication (including herbal remedies) during the two weeks before the start of the study or OTC medicinal products (including herbal remedies) during the week before study initiation and throughout the study;
9. Use of medications such as benzodiazepines, anticonvulsants, or barbiturates for one month before the start of the study and throughout the study;
10. Trial participant consumed tobacco/tobacco-containing products, pan or pan masala, gutkha, and masala (containing beetle nut and tobacco) for at least 48.00 hours before initiation of the study and throughout the study;
11. Trial participant consumed caffeine and/or xanthine-containing foods or beverages (i.e., coffee, tea, chocolate, and caffeine-containing sodas, colas, etc.) and grapefruit juice and poppy-containing foods for at least 48.00 hours before initiation of the study and throughout the study;
12. Major illness during the 90 days before screening;
13. Participation in a drug research study within 90 days of screening;
14. Positive screening test result for any one or more of the following: HIV, Hepatitis B, Hepatitis C, and VDRL;
15. History or presence of easy bruising or bleeding;
16. Abnormal diet pattern for whatever reason (e.g., low sodium, fasting, and high protein diets) during the four weeks preceding the study;
17. Females of childbearing potential with any one of the following reported and documented on the medical history:

    i.Postmenopausal with spontaneous amenorrhea for at least one year, or ii.Bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or iii.Total hysterectomy and an absence of bleeding for at least 3 months; iv.Female volunteers who have used implanted or injected hormonal contraceptives anytime during the 6 months prior to study or used hormonal contraceptives within 07 days before dosing;
18. Pregnant women and nursing mothers;
19. Male and females of childbearing potential unwilling to employ appropriate and reliable method of contraception like non-hormonal intrauterine devices, barrier methods, and spermicidal agents, Double Barrier method (Condom) during the study till 07 days after the completion of the study;
20. Male volunteers willing to donate sperm during the study till 07 days after the completion of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of Urolithin A over time and maximal plasma concentration (Cmax) | Pharmacokinetic blood samples will be collected at pre-dose [within 45 min before product administration] and post-dose at 1-hours; 4-hours; 6-hours; 8-hours; 12-hours; 24-hours; and 72-hours. (Total 08 Time points).
Exposure to Urolithin A over time measured as area under the curve (AUC) | 72-hours

SECONDARY OUTCOMES:
Number of adverse events and serious adverse events throughout the study. | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ramshyam Agarwal, MD, Principal Investigator — Lokmanya Medical Research Centre and Hospital
Locations (1):
- Lokmanya Medical Research Centre and Hospital, Pune, India

IPD SHARING:
Plan to Share IPD: No